CLINICAL TRIAL: NCT02768155
Title: Protocol for the Clinical Evaluation Amniotic Fluid (AF) Product in Knee Osteoarthritis
Brief Title: Evaluation of Amniotic Fluid Product in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OFORT001
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis of the Knee
Keywords: OA, Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AF 4.0 (Experimental): Amniotic Fluid 4.0ml dose
  Interventions: Other: Amniotic Fluid 4.0ml dose
- AF 2.0 (Experimental): Amniotic Fluid 2.0ml dose
  Interventions: Other: Amniotic Fluid 2.0ml dose
- Placebo (Placebo Comparator): Saline Placebo Control
  Interventions: Other: Placebo Control

INTERVENTIONS:
Other: Amniotic Fluid 4.0ml dose — Injection of Amniotic Fluid
  Arms: AF 4.0
Other: Amniotic Fluid 2.0ml dose — Injection of Amniotic Fluid
  Arms: AF 2.0
Other: Placebo Control — Normal Saline
  Arms: Placebo

SUMMARY:
A study evaluating Amniotic Fluid compared to a Saline Placebo Injection in the treatment of subjects with osteoarthritic (OA) knee pain

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 30 years or older.
2. Subject has a diagnosis of osteoarthritis (OA) defined as Grade 1 to 3 on the Kellgren Lawrence grading scale.
3. Subject is willing and able provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study.

Exclusion Criteria:

1. Subject has active infection at the injection site.
2. Subject has rheumatoid arthritis, psoriatic arthritis, or have been diagnosed with any other auto-immune disorders that could be the cause of their knee pain.
3. BMI greater than 45 kg/m2
4. Subject has received an intra-articular hyaluronic acid (HA) injection for the treatment of OA of the target knee within 3 months prior to screening.
5. Subject has received a steroid or platelet rich plasma (PRP) injection for the treatment of OA of the target knee within 3 months prior to screening.
6. Subject has had major surgery, arthroplasty or arthroscopy in the target knee within 26 weeks of treatment or plans to have surgery in the target knee within 180 days of treatment.
7. Subject is pregnant or plans to become pregnant within 180 days of treatment.
8. Subject has used an investigational drug, device or biologic within 12 weeks prior to treatment.
9. Subject has any significant medical condition that, in the opinion of the Investigator, would interfere with protocol evaluation and participation.
10. Subject has a history of immunosuppressive or chemotherapy in the last 5 years
11. Subject has autoimmune disease or a known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV
12. Subject has had prior radiation at the site
13. Subject is currently taking anticoagulant therapy (excluding Plavix or Aspirin)
14. Diagnosis of gout in the past 6 month
15. Subject has a diagnosis of osteoarthritis

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Reduction in Pain | 3 months

SECONDARY OUTCOMES:
Range of Motion | 3 month
Knee injury and Osteoarthritis Outcome Score (KOOS) | 3 month
WOMAC | 3 month
Kellgren-Lawrence grade of OA | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald Fetterolf, MD, Study Director — MiMedx Group, Inc.
Locations (2):
- United States (2):
  - Central Research Associates, Inc, Birmingham, Alabama
  - Weil Foot, Ankle and Orthopedic Institute, Des Plaines, Illinois

IPD SHARING:
Plan to Share IPD: No